CLINICAL TRIAL: NCT00971464
Title: A Randomized Controlled Trial of Eccentric Viewing Training vs. Closed Circuit Television Use for Visual Rehabilitation From Age-Related Macular Degeneration
Brief Title: Low Vision Study Comparing EV Training vs. CCTV for AMD Rehabilitation
Acronym: AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, William Hodge, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-08-683; 15968E (Other: REB)
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: AMD
Keywords: AMD; EV; CCTV; Reading; vision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric viewing (Experimental): Eccentric viewing is the use of a retinal locus other than the anatomical fovea for fixation in cases when there is central vision loss. This other area (or areas) is called the preferred retinal locus (PRL). In eccentric viewing the patient is aware that they are "looking to the side" or "using their side vision". Most patients with a dense central scotoma will develop eccentric viewing naturally over time. It is thought, however, that, in many cases the naturally developed PRL is not in the ideal position. The four components of eccentric viewing that will be taught are: 1) The optimal direction for eccentric viewing 2) Using large objects to teach eccentric viewing 3) Repetitive practicing of the technique and 4) Maintaining the eye in the eccentric viewing position.
  Interventions: Behavioral: eccentric viewing (EV) training
- CCTV arm (Active Comparator): A CCTV is an electro-optical device mainly used for reading, but which can also be used for writing or viewing pictures. It is comprised of a video camera which faces downwards towards the reading material and which inputs the image to a digital monitor. Magnification is variable over a large range. By means of a zoom lens and the brightness, contrast, and image polarity (black letters on white or white on black) can be controlled to provide the best combination of viewing conditions for an individual user. The significant advantages of CCTV over optical magnifiers are that it provides high levels of magnification with a greater field of view (compared to the equivalent optical device), allows reading at a more normal viewing distance of about 40 - 50 cms and allows binocular viewing.
  Interventions: Device: Closed circuit television (CCTV)

INTERVENTIONS:
Behavioral: eccentric viewing (EV) training — Eccentric viewing training for 6 weeks, minimum two 10 minutes per day.
  Other Names: eccentric fixation training, vision training
  Arms: Eccentric viewing
Device: Closed circuit television (CCTV) — A CCTV is an electro-optical device mainly used for reading.
  Other Names: EVES, electronic vision enhancement system
  Arms: CCTV arm

SUMMARY:
Patients with advanced Age-Related Macular Degeneration will be randomized into one of two treatment groups. One group will receive eccentric view (EV) training while the other a closed circuit television (CCTV) training for 6 weeks. Reading speed and accuracy will be assessed pre- and post- treatment to determine if one treatment is superior to the other.

DETAILED DESCRIPTION:
Age-related macular degeneration is the single most common cause of visual impairment in Canada, affecting people over the age of 55 years. It causes loss of central, detailed vision, resulting in difficulty with fine vision tasks, such as reading and writing. At present there is no fully effective prevention or treatment for this condition, but people do benefit from visual rehabilitation. Two of the most common rehabilitation techniques are eccentric viewing training and an electronic magnification system called a Closed circuit television (CCTV). In eccentric viewing training the person is taught to use his or her remaining side vision, instead of central vision. The CCTV provides high levels of magnification to compensate for the loss of detail vision. The purpose of this randomized clinical trial is to compare the effectiveness of these two interventions. In the study people will be randomly assigned to either receiving eccentric viewing training or a CCTV. This will happen after they have received basic, optical low vision services and training through the CNIB. We will assess their performance with either the CCTV or EV training with a variety of reading tasks and questionnaires. The results will give evidence for how it is most beneficial to use resources and as such will be very important in future planning of low vision services.

Hypothesis: Eccentric Viewing Training will improve reading speed over CCTV by at least 10 words per minute in patients with advanced AMD.

ELIGIBILITY:
Inclusion Criteria:

* First time AMD patient sent to CNIB for visual rehabilitation
* Macular Degeneration reducing visual acuity (VA) to between 20/160 and 20/400 (ETDRS scale)
* Over the age of 50 years
* English as the first language and able to read

Exclusion Criteria:

* Expected anti-VEGF or Visudyne treatment over the course of the study
* Individuals who do not have reading as a life goal
* Mental cognition that makes learning the specific rehabilitation tasks unlikely (determined by mini-mental state exam)
* Any other ocular pathology that can reduce central vision including cornea decompensation (scar or thickness), cataract (grade III or more for each type of cataract), vitritis (2+ or more) or advanced glaucoma (C/D ratio of >0.7)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures reading speed for 1.3M print (in correct words per minute). | 6 weeks intervention

SECONDARY OUTCOMES:
The secondary outcomes measures 1. Reading accuracy for 1.3M; | 6 weeks intervention
2. Reading speed and accuracy for 1M | 6 weeks intervention
3. Reading performance tests. | 6 week's intervention
4. Reading Behavior Inventory | 6 week's intervention
5. VFQ-25 plus 2 extra questions). | 6 week's intervention
6. Geriatric depression scale | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: William Hodge, MD, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- CNIB, Toronto Branch, Toronto, Ontario, Canada